CLINICAL TRIAL: NCT02792127
Title: Online Cognitive Behavioural Therapy Program for Social Anxiety
Brief Title: Online Program for Social Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Frances Chen, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: H16-00319
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Social Anxiety
Keywords: Social Anxiety; Cognitive Behaviour Therapy; Online Program

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): These participants will be given access to a six-month online program for social anxiety.
  Interventions: Behavioral: Online Program for Social Anxiety
- Wait List Control (No Intervention): These participants will not be given an intervention until after they have completed the study.

INTERVENTIONS:
Behavioral: Online Program for Social Anxiety — This program will be completed from participants' homes using their own computers. This online format is based on a Cognitive Behaviour Therapy framework (CBT) and involves seven modules that ask participants to engage in a variety of thinking exercises and activities.
  Arms: Experimental

SUMMARY:
The purpose of this study is to investigate the efficacy of an online program in reducing symptoms of social anxiety, unhelpful thoughts, avoidance behaviours, fear of negative evaluations and improving quality of life in students with above-average social anxiety.

DETAILED DESCRIPTION:
While there are many benefits to online programs in treating a variety of health issues (i.e., implementation in remote areas, cost-effectiveness, etc.), the primary challenge for online formats is to imitate real-life interactions while promoting a reduction in symptoms. This will be attempted in a six-month online program for social anxiety.

The present study will assess the efficacy of a six-month online program through measures of social anxiety, fear of negative evaluations, unhelpful thoughts, avoidance behaviours and quality of life. This information will be collected from students at baseline and upon completion of the online program.

ELIGIBILITY:
Inclusion Criteria:

* Registered UBC student
* Achieve an above-average score on a validated screening tool for social anxiety

Exclusion Criteria:

* Not a registered UBC student
* Clinical diagnosis of a mental illness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-07; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Social Anxiety | six months
  A self-report measure that assesses symptoms of distress experienced when socializing with others.

CONTACTS AND LOCATIONS:
Overall Officials: Frances Chen, PhD, Principal Investigator — University of British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Helgadottir FD, Ross MG, Onslow M, Packman A, O'Brian, S. Online CBT II: A phase I trial of a standalone, online CBT Treatment Program for Social Anxiety in Stuttering. Behaviour Change 26(4): 254-270. 2009.
- [Background] Helgadottir FD, Menzies RG, Onslow M, Packman A, O'Brian S. Online CBT I: Bridging the gap between Eliza and modern online CBT treatment packages. Behaviour Change 26(4): 245-253, 2009.
- [Derived] McCall HC, Richardson CG, Helgadottir FD, Chen FS. Evaluating a Web-Based Social Anxiety Intervention Among University Students: Randomized Controlled Trial. J Med Internet Res. 2018 Mar 21;20(3):e91. doi: 10.2196/jmir.8630. PMID 29563078